CLINICAL TRIAL: NCT06788184
Title: Development and Evaluation of the Effectiveness of a Virtual Reality Game Targeting Central Auditory Processing Skills in Children Using Cochlear Implants
Brief Title: Virtual Reality Game to Enhance Auditory Processing in Children With Cochlear Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Seyma Nur TABAK, Research Assistant, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37/2024; Scientific Research Projects (Other: Istanbul Aydin University Scientific Research Projects)
Record Dates: First submitted 2025-01-12; First posted 2025-01-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Central Auditory Processing Disorder
Keywords: Cochlear Implant; Auditory Processing; Virtual Reality; Auditory Attention; Working Memory
MeSH Terms: conditions — Language Development Disorders | interventions — Auscultation

STUDY DESIGN:
Intervention Model Description: This interventional study adopts a parallel group design, comparing the effects of a virtual reality (VR)-based auditory rehabilitation program with traditional auditory rehabilitation methods in children aged 10-18 years who use bilateral cochlear implants. Participants will be randomly assigned to two groups:
  Intervention Group: Participants in this group will engage in a virtual reality game designed to enhance central auditory processing skills. The VR game includes tasks focusing on auditory attention, working memory, auditory localization, and speech perception in noise. The intervention will consist of weekly 30-minute sessions over a 4-week period.
  Control Group: Participants in this group will undergo traditional auditory rehabilitation, following established methods aimed at improving similar auditory processing skills.
  The study model ensures a structured comparison of the effectiveness of the VR intervention against conventional methods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Traditional Auditory Rehabilitation Only) (Active Comparator): Participants in the control group (15 bilateral cochlear implant users, aged 10-18 years) will receive traditional auditory rehabilitation sessions once a week for 30 minutes over a 4-week period. This group will not participate in the virtual reality intervention.
  Interventions: Behavioral: Traditional Auditory Rehabilitation
- Experimental Group (Traditional Auditory Rehabilitation + VR Game) (Active Comparator): This group will include 15 participants aged 10-18 years with bilateral cochlear implants. In addition to traditional auditory rehabilitation, participants will receive virtual reality (VR) game-based rehabilitation for 30 minutes once a week. The intervention will last for 4 weeks and aims to improve central auditory processing skills.
  Interventions: Device: Virtual Reality (VR) Game for Auditory Processing; Behavioral: Traditional Auditory Rehabilitation

INTERVENTIONS:
Device: Virtual Reality (VR) Game for Auditory Processing — The Virtual Reality (VR) Game is a novel auditory rehabilitation tool designed to enhance central auditory processing skills in children with cochlear implants. This intervention features a restaurant simulation environment where participants perform auditory tasks such as identifying verbal orders, recognizing speech in noisy environments, and matching auditory cues to visual inputs.
  Dosage Form: Virtual reality sessions conducted through a VR headset (Oculus Meta Quest 3).
  Frequency: Once per week. Duration per Session: 30 minutes per session. Total Duration: Four weeks (4 sessions). Complexity Levels: Tasks increase in complexity over time, starting with simple auditory cues in quiet environments and progressing to more challenging scenarios involving background noise and multitasking.
  The VR game is specifically designed to replicate real-world auditory challenges in a controlled and engaging virtual environment, providing participants with tailored tasks to improve auditory atten
  Arms: Experimental Group (Traditional Auditory Rehabilitation + VR Game)
Behavioral: Traditional Auditory Rehabilitation — Name: Traditional Auditory Rehabilitation
  Description:
  Participants will continue the standard auditory rehabilitation program they currently receive at their registered rehabilitation center and will focus on improving auditory processing skills. This program includes:
  Session Length: 30 minutes per session Frequency: Once a week Total Duration: 4 weeks (4 sessions total)
  Components:
  Improve speech understanding in noise

SUMMARY:
This study aimed to design and evaluate the effectiveness of a virtual reality-based restaurant simulation game to improve central auditory processing skills in children with bilateral cochlear implants. The study aims to improve auditory attention, working memory, and speech perception in noise. Children with bilateral cochlear implants between the ages of 10 and 18 will participate in this study, which combines traditional rehabilitation methods with a virtual reality game. The "Hearing in Noise Test" (HINT) assessment tools will be used. The game aims to present interactive scenarios that simulate auditory difficulties encountered in daily life and to improve auditory processing skills. The usability of the game will be tested in the pilot phase. This project aims to bring an innovative approach to rehabilitation programs and to contribute to the social integration of children with hearing loss while increasing social awareness.

DETAILED DESCRIPTION:
This study aims to develop and evaluate a virtual reality (VR) game designed to improve central auditory processing skills in children aged 10-18 years with bilateral cochlear implants. The project aims to test the effectiveness of an innovative VR platform as a complement to traditional auditory rehabilitation methods. It focuses on improving critical skills such as auditory attention in noise, working memory, auditory localization and speech perception.

Scope of the Study:

Participant Profile: Children aged 10-18 years with prelingual hearing loss who received bilateral cochlear implants before the age of 2. Participants will be selected according to the criteria of the Child Auditory Performance Scale (CHAPS) and a minimum age of 7 years for receptive and expressive language as a result of the Peabody Picture Word Test.

Methodology: The study will compare traditional auditory rehabilitation (control group) with VR-based rehabilitation (study group). The VR rehabilitation process will consist of weekly 30-minute sessions lasting a total of 4 weeks. The assessment tools will include the Hearing in Noise Test (HINT).

Scales and Forms to be Used in the Pilot Study: The following tools and forms will be used in the pilot phase to comprehensively evaluate the effectiveness and usability of the game:

Demographic Information Forms:

Demographic information form for children using cochlear implants. Demographic information form for children with normal hearing. Game Observation Checklist: Used to systematically observe and document participants' interactions with the game.

Virtual Reality Game Test List: To evaluate specific tasks and performance results in the VR game.

System Usability Scale (SUS): Will be administered to parents to evaluate the usability of the VR system. Parents will provide insight into how their children experienced the game and their perceptions of the usability process.

Parent One-on-One Interview Form: To collect feedback from parents about the impact and effectiveness of the game. Child Game Evaluation Form: To collect direct feedback from children about their experiences with the VR game.

Participant One-on-One Interview Form: To document qualitative data from participants about their experiences and challenges.

The feedback received from 10 participants and their parents in the pilot phase will play a critical role in improving the game mechanics and ensuring the effectiveness of the system.

Innovative Aspects and Contributions: The innovative aspect of the study is the use of virtual reality technology in auditory rehabilitation. In the VR environment, participants will undertake tasks in a realistic restaurant simulation by adapting to increasing levels of difficulty to improve their auditory skills. The study aims to achieve improvements in auditory attention, working memory and speech perception in noise of the participants, exceeding the results of traditional methods.

It is expected that the results of this study will contribute to the development of new strategies for the rehabilitation of individuals with hearing loss and enable them to participate more effectively in daily life. In addition, the developed VR game will support the education and social integration of hearing impaired individuals while raising awareness in society. It is planned that the scientific findings of the study will be published in national and international journals and form the basis for the development of various rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Being between 10 and 18 years old
* Having bilateral cochlear implants
* Having prelingual hearing loss before the age of 2 and having a cochlear implant
* Having a minimum receptive and expressive language age of 7 on the Peabody Picture-Word Test
* Having no additional condition that may cause dizziness or balance disorders
* Having a score in the following ranges on the Child Hearing Performance Scale (CHAPS):

  * Noise Environment item: -7 to -21
  * Multiple Stimuli item: -3 to -9
  * Auditory Memory item: -8 to -24
  * Auditory Attention Span item: -8 to -24
* Having no diagnosed neurodevelopmental disorder
* Being a native Turkish speaker
* Being willing to participate in the study and signing the informed consent form.

Exclusion Criteria:

* Individuals younger than 10 or older than 18 years old.
* Individuals using unilateral cochlear implants.
* Individuals without prelingual hearing loss or who had a cochlear implant after the age of 2.
* Individuals with a receptive and expressive language age of under 7 as a result of the Peabody Picture-Word Test.
* Individuals with dizziness, balance disorders or neurodevelopmental problems.
* According to the results of the Child Auditory Performance Scale (CHAPS):

  * Those who scored under -7 or over -21 on the "Noise" subscale.
  * Those who scored under -3 or over -9 on the "Multiple Input" subscale.
  * Those who scored under -8 or over -24 on the "Auditory Memory" subscale.
  * Those who scored under -8 or over -24 on the "Auditory Attention Span" subscale.
* Individuals whose native language is not Turkish.
* Individuals who did not want to participate in the study and/or did not sign the informed consent form.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Speech Recognition in Noise Using the Hearing in Noise Test (HINT) | The outcome will be assessed at Baseline (Week 0) and Post-Intervention (Week 4), with improvements in scores reflecting better speech perception in noise.
  The HINT test is an adaptable test for measuring sentence recognition threshold, which evaluates the status and efficiency of hearing in noise using sentences from daily life. The aim of the HINT test is to evaluate the auditory capacity of the individual in noisy environments.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydın University, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared to ensure the privacy and confidentiality of the participants. As the study involves a vulnerable group of children with cochlear implants, maintaining their personal data's integrity is of utmost importance. Additionally, the ethical committee's guidelines and institutional policies require strict data protection to prevent potential misuse. Therefore, the IPD will remain confidential and will not be made publicly available.

REFERENCES:
- [Derived] Tabak SN, Meral Cetinkaya M, Irali AE. Development and evaluation of a virtual reality game targeting Central auditory processing skills in children using cochlear implants: a randomized controlled trial. Disabil Rehabil Assist Technol. 2026 Feb 4:1-18. doi: 10.1080/17483107.2026.2623465. Online ahead of print. PMID 41636301